CLINICAL TRIAL: NCT04016259
Title: Self Cranial Electrical Stimulation for Pain in Older Adults With Knee Osteoarthritis (Self CES for Knee Pain)
Brief Title: Self Cranial Electrical Stimulation (CES) for Pain in Older Adults With Knee Osteoarthritis (Self CES for Knee Pain)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Hyochol Ahn, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-SN-19-0452
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Self-CES (Experimental)
  Interventions: Device: Cranial Electrical Stimulation (CES)
- Sham-CES (Placebo Comparator)
  Interventions: Device: Sham-CES

INTERVENTIONS:
Device: Cranial Electrical Stimulation (CES) — CES will be applied for 60 minutes per session daily for 2 weeks (Monday to Friday) via the Alpha-Stim M Electromedical Products International, Inc., Mineral Wells, TX).
  Other Names: Alpha-Stim M
  Arms: Self-CES
Device: Sham-CES — For sham CES, the electrodes will be identical look and be placed in the same positions as for active stimulation, but the stimulator will not deliver electrical current.
  Other Names: Alpha-Stim M
  Arms: Sham-CES

SUMMARY:
The purpose of this study is to determine the feasibility, safety, and preliminary efficacy of a two-week self Cranial Electrical Stimulation(CES) on pain in older adults with knee osteoarthritis(OA)

ELIGIBILITY:
Inclusion Criteria:

* have self-reported unilateral or bilateral knee OA pain, according to American College of Rheumatology criteria
* have had knee OA pain in the past 3 months with an average of at least 30 on a 100 Numeric Rating Scale (NRS) for pain
* can speak and read English
* have a device with internet access that can be used for secure video conferencing for real- time remote supervision
* have no plan to change medication regimens for pain throughout the trial
* are able to travel to the coordinating center
* are willing and able to provide written informed consent prior to enrollment

Exclusion Criteria:

* history of brain surgery, brain tumor, seizure,stroke, or intracranial metal implantation
* serious medical illness, such as uncontrolled hypertension (i.e., systolic blood pressure/ diastolic blood pressure ≥ 150/95 mm Hg)heart failure, or history of acute myocardial infarction
* alcohol/substance abuse
* cognitive impairment
* pregnancy or lactation
* hospitalization within the preceding year for psychiatric illness

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyochol Ahn, PhD, RN, MSN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham-CES | Self-CES
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham-CES | Self-CES | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.13 (5.83) | 59.77 (6.88) | 59.43 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 2
  White | 7 | 8 | 15
  African American | 5 | 3 | 8
  Hispanic | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Education [Count of Participants; unit: Participants]
  < High school | 5 | 6 | 11
  2-Year College | 1 | 4 | 5
  4-Year College | 5 | 2 | 7
  Master's Degree | 3 | 2 | 5
  Doctoral Degree | 1 | 1 | 2
Duration of Osteoarthritis [Mean (Standard Deviation); unit: months] | 55.87 (40.64) | 108 (103.87) | 81.03 (80.86)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.66 (8.33) | 32.56 (8.17) | 33.11 (8.13)
Pain as Assessed by a Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — The NRS total score ranges from 0 (no pain) to 100 (most intense pain imaginable).
  units on a scale | 34.67 (32.48) | 44.33 (19.90) | 39.50 (26.92)
Clinical pain assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) [Mean (Standard Deviation); unit: score on a scale] — The WOMAC ranges from 0 to 96, with higher scores indicating worse osteoarthritis (OA) pain-related symptoms
  score on a scale | 52.67 (21.413) | 52.20 (17.604) | 52.44 (19.5085)
Experimental Pain Sensitivity as measured by heat pain threshold (HPTH) [Mean (Standard Deviation); unit: degree Celsius] — In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  degree Celsius | 40.12 (2.69) | 38.34 (3.44) | 39.23 (3.16)
Experimental Pain Sensitivity as measured by heat pain tolerance (HPTO) [Mean (Standard Deviation); unit: degree Celsius] — In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  degree Celsius | 43.85 (3.26) | 43.22 (3.15) | 43.54 (3.16)
Experimental Pain Sensitivity as measured by pressure pain threshold (PPT) [Mean (Standard Deviation); unit: kilogram-force (kgf)] — In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  kilogram-force (kgf) | 1.86 (1.32) | 1.60 (0.95) | 1.73 (1.14)
Experimental Pain Sensitivity as measured by Conditioned Pain Modulation (CPM) [Mean (Standard Deviation); unit: kilogram-force (kgf)] — In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  kilogram-force (kgf) | 2.70 (1.26) | 2.53 (0.86) | 2.61 (1.06)
Psychosocial symptoms measured by the Patient-Reported Outcomes Measurement Info System - anxiety [Mean (Standard Deviation); unit: score on a scale] — The 7-item Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form assesses the pure domain of anxiety in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
  score on a scale | 15.67 (8.723) | 12.27 (4.200) | 13.97 (6.4615)
Psychosocial symptoms as measured by PROMIS - depression [Mean (Standard Deviation); unit: score on a scale] — The 8-item PROMIS Depression Short Form assesses the pure domain of depression in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
  score on a scale | 12.73 (5.351) | 10.53 (2.446) | 11.63 (3.8985)
Psychosocial symptoms as measured by PROMIS - sleep disturbance [Mean (Standard Deviation); unit: score on a scale] — The 8-item PROMIS Sleep Disturbance Short Form assesses the pure domain of sleep disturbance in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely;3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
  score on a scale | 27.47 (7.029) | 22.20 (8.187) | 24.835 (7.608)
Psychosocial symptoms as measured by the Pain Catastrophizing Scale (PCS) [Mean (Standard Deviation); unit: score on a scale] — The Pain Catastrophizing Scale (PCS) consists of 13 items assessing three components of catastrophizing: rumination, magnification, and helplessness. It is measured using the 0 (not at all) to 4 (all the time) scale. Total score ranges from 0 to 52, with higher scores indicating greater pain catastrophizing.
  score on a scale | 18.40 (14.495) | 13.80 (10.065) | 16.10 (12.280)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pain as Assessed by a Numeric Rating Scale (NRS) for Pain
Description: The NRS total score ranges from 0 (no pain) to 100 (most intense pain imaginable).
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
units on a scale | 40.40 (33.79) | 27.33 (16.89)

2. Primary Outcome: Clinical Pain as Assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The WOMAC ranges from 0 to 96, with higher scores indicating worse osteoarthritis (OA) pain-related symptoms
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
score on a scale | 47.40 (25.136) | 43.80 (18.040)

3. Secondary Outcome: Experimental Pain Sensitivity as Measured Using a Multimodal Quantitative Sensory Testing (QST) Battery - Heat Pain Threshold (HPTH)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  To assess HPTH, heat stimuli were delivered to the participant's knee using a computer-controlled TSAII NeuroSensory Analyzer. From a baseline of 32 degrees Celsius, the temperature increased by 0.5 degrees Celsius per second until the participants responded by pressing a button to stop heat stimuli. Participants were instructed to press the button when the sensation ''first becomes painful" to assess the heat pain threshold (HPTH).
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
degree Celsius | 37.90 (2.03) | 41.04 (3.17)

4. Secondary Outcome: Experimental Pain Sensitivity as Measured Using a Multimodal Quantitative Sensory Testing (QST) Battery - Heat Pain Tolerance (HPTO)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  To assess HPTO, heat stimuli were delivered to the participant's knee using a computer-controlled TSAII NeuroSensory Analyzer. From a baseline of 32 degrees Celsius, the temperature increased by 0.5 degrees Celsius per second until the participants responded by pressing a button to stop heat stimuli. Participants were instructed to press the button when they ''no longer feel able to tolerate the pain" to assess their heat pain tolerance (HPTO).
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
degree Celsius | 43.05 (2.77) | 44.56 (3.12)

5. Secondary Outcome: Experimental Pain Sensitivity as Measured Using a Multimodal Quantitative Sensory Testing (QST) Battery - Pressure Pain Threshold (PPT)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  To assess PPT, a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's knee. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful" to assess pressure pain threshold (PPT).
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
kilograms force (kgf) | 1.06 (0.48) | 2.59 (1.46)

6. Secondary Outcome: Experimental Pain Sensitivity as Measured Using a Multimodal Quantitative Sensory Testing (QST) Battery - Conditioned Pain Modulation (CPM)
Description: In order to measure experimental pain sensitivity, a multimodal Quantitative Sensory Testing (QST) battery will be completed: heat pain threshold (HPTH), heat pain tolerance (HPTO), pressure pain threshold (PPT), and Conditioned Pain Modulation (CPM).
  CPM was assessed as the change in PPT on the trapezius immediately after the immersion of the contralateral hand up to the wrist in a cold-water bath (Neslab, Portsmouth, NH) at 12 degrees C for one minute. [To assess PPT, a handheld digital pressure algometer (Wagner, Greenwich, CT) was applied at a constant rate of 0.3 kilograms force per centimeter squared (kgf/cm^2) per second to the participant's trapezius. Participants were asked to notify the experimenter when the pressure sensation ''first becomes painful" to assess pressure pain threshold (PPT).]
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: kilograms force (kgf)
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
kilograms force (kgf) | 1.93 (0.90) | 3.64 (1.67)

7. Secondary Outcome: Psychosocial Symptoms as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety Short Form
Description: The 7-item PROMIS Anxiety Short Form assesses the pure domain of anxiety in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
score on a scale | 15.13 (6.770) | 13.20 (4.663)

8. Secondary Outcome: Psychosocial Symptoms as Measured by PROMIS - Depression Short Form
Description: The 8-item PROMIS Depression Short Form assesses the pure domain of depression in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression.
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
score on a scale | 13.13 (5.449) | 10.87 (2.642)

9. Secondary Outcome: Psychosocial Symptoms as Measured by PROMIS - Sleep Disturbance Short Form
Description: The 8-item PROMIS Sleep Disturbance Short Form assesses the pure domain of sleep disturbance in individuals age 18 and older, and each item on the measure is rated on a 5-point scale (1=never; 2=rarely;3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
score on a scale | 24.60 (6.566) | 22.27 (7.126)

10. Secondary Outcome: Psychosocial Symptoms as Measured by the Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) consists of 13 items assessing three components of catastrophizing: rumination, magnification, and helplessness. It is measured using the 0 (not at all) to 4 (all the time) scale. Total score ranges from 0 to 52, with higher scores indicating greater pain catastrophizing.
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
score on a scale | 15.87 (15.505) | 14.47 (10.789)

11. Secondary Outcome: Number of Participants With a Significant Change in Pain-related Cortical Response on Average as Assessed by a Continuous Wave, Multichannel Functional Near-infrared Spectroscopy (fNIRS) Imaging System
Description: Pain-related cortical response will be measured using a continuous-wave, multichannel fNIRS imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan) with three semiconductor lasers at 780, 805, and 830 nm. Optical recordings will be collected during thermal pain stimulation.
Time Frame: baseline, week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
Participants | 0 | 15

12. Secondary Outcome: Participant Satisfaction With Treatment Using the Client Satisfaction Questionnaire (CSQ-8)
Description: The CSQ-8 comprises eight items that are summed to yield an overall score of 8-32, with higher scores indicating greater satisfaction.
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
score on a scale | 29.53 (2.264) | 27.20 (4.843)

13. Secondary Outcome: Feasibility as Measured by the Number of Participants That Completed the Full CES Protocol
Time Frame: week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

14. Secondary Outcome: Feasibility as Indicated by Participant's Cranial Electrical Stimulation (CES) Experience
Description: CES experience will be measured on a 10-item scale, with each item rated 0-10 and 0 being strongly disagree and 10 being strongly agree. Total score ranges from 0 to 100, with higher scores indicating a better CES experience.
  Question 1. It was easy to prepare the device and accessories Question 2. The device was unnecessarily complex Question 3. The device was easy to use Question 4. I felt the video conferences with a technical person were helpful Question 5. I would imagine that most people would learn to use this device quickly Question 6. The device was cumbersome to use Question 7. I felt confident using the device Question 8. I needed to learn a lot of things before I could get going with this device Question 9. The effectiveness of the treatment increased over the course of treatment Question 10. I felt that transcranial electrical stimulation treatment benefited me
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
units on a scale
  Question 1 | 9.80 (0.56) | 9.93 (0.26)
  Question 2 | 0.00 (0.00) | 0.00 (0.00)
  Question 3 | 9.93 (0.29) | 10.00 (0.00)
  Question 4 | 8.73 (2.55) | 9.27 (1.94)
  Question 5 | 9.67 (0.62) | 9.87 (0.52)
  Question 6 | 0.27 (0.70) | 0.07 (0.26)
  Question 7 | 9.67 (1.29) | 10.00 (0.00)
  Question 8 | 0.53 (1.36) | 0.20 (0.56)
  Question 9 | 6.47 (3.50) | 5.67 (4.35)
  Question 10 | 5.80 (3.55) | 6.33 (4.10)

15. Secondary Outcome: Tolerability as Indicated by Number of Participants With Possible Side Effects of Treatment
Description: Measurement of presence and severity of possible side effects of treatment on a 0 (not at all) to 10 (highest degree) scale.If any side effects are reported, the degree of relatedness to the intervention will be assessed on a 5-point scale.
Time Frame: week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sham-CES | Self-CES
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Sham-CES | Self-CES
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Small sample size; limited demographic (older adults with knee OA) restricts generalizability; slight deviations among intervals between daily stimulation sessions (though, this may be consistent with real-world use); long term efficacy not evaluated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT04016259/Prot_SAP_000.pdf